CLINICAL TRIAL: NCT06973252
Title: The Effect of Eye Mask on Sleep Quality in Patients Hospitalised in Surgical Intensive Care Unit: Non-Randomised Experimental Study
Brief Title: Sleep Quality in Surgical Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, PhD, Research Assisstant (Principal Investigator), Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sleep Quality
Record Dates: First submitted 2025-05-14; First posted 2025-05-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Nursing Care; Intensive Care Unit ICU; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group patients were fitted with an eye mask designed by the researcher by placing a black fabric in the size of the mask between two three-layer surgical masks with Asfor brand soft elastic earphones and stapling the edges. The designed eye mask was cut with scissors according to the shape of the nose so that the mask would fit the eye exactly and prevent the light from entering the eye. A separate mask was used for each patient in the intervention group. Patients who were admitted to the SICU after surgery were evaluated for agitation-pain-delirium at 23:00 on postoperative days 0, 1, and 2, were told to wear their eye masks after the scale application, and the patients were allowed to sleep at 23:00 at the latest. Patients were allowed to remove the eye patch for short periods of time (10 minutes or less at a time) and then put it back on when uncomfortable and when necessary.
  Interventions: Behavioral: Eye masks
- Control group (No Intervention): Control group received the usual care.

INTERVENTIONS:
Behavioral: Eye masks — The intervention group patients were fitted with an eye mask designed by the researcher by placing a black fabric in the size of the mask between two three-layer surgical masks with Asfor brand soft elastic earphones and stapling the edges. The designed eye mask was cut with scissors according to the shape of the nose so that the mask would fit the eye exactly and prevent the light from entering the eye. A separate mask was used for each patient in the intervention group. Patients who were admitted to the NICU after surgery were evaluated for agitation-pain-delirium at 23:00 on postoperative days 0, 1, and 2, were told to wear their eye masks after the scale application, and the patients were allowed to sleep at 23:00 at the latest. Patients were allowed to remove the eye patch for short periods of time (10 minutes or less at a time) and then put it back on when uncomfortable and when necessary.
  Arms: Intervention group

SUMMARY:
It is thought that transferring low-cost and easily applicable interventions that can be used to control environmental stressors such as noise and light that negatively affect sleep quality, especially in intensive care environments, into clinical practice will improve the quality of nursing care. It is recommended that complementary interventions that can be used to improve such sleep quality should be tested and supported by new studies. In this study, it was aimed to determine the effect of eye mask on sleep quality in patients admitted to the surgical intensive care unit after abdominal surgery.

DETAILED DESCRIPTION:
Sleep is one of the basic needs to maintain and protect health and is a physiological state that occurs as a result of loss of consciousness, slowing of muscle activities, and decrease in neural activity for a certain period of time. Sleep quality is adversely affected as a result of physiological or psychological factors occurring in the perioperative period or disruptions in normal sleep phases due to environmental factors such as light and noise in the intensive care environment. Especially in surgical intensive care units (SICU), it is one of the units where deterioration in the sleep quality of patients is frequently experienced.

It is reported that improving sleep quality in intensive care units will support the recovery processes of patients in the clinical environment and shorten the duration of hospital stay. Non-pharmacological methods are frequently used in patients hospitalised in the intensive care unit. In the literature, there are research results on the positive effects of using eye patch and earplugs, listening to audio books, massage and aromatherapy, acupressure, music therapy, white noise application, reflexology massage and foot bath interventions on sleep quality.

Sleep is an important component of nursing management in surgical intensive care units and is one of the basic needs of patients. Surgical nurses who provide nursing care here should plan, implement and evaluate environmental arrangements and non-pharmacological interventions to improve the sleep quality of patients. Especially interventions such as eye mask can be used to control the environmental factor that negatively affects sleep quality in surgical intensive care units. In systematic reviews and meta-analyses on the method of sleep in intensive care unit patients, it is reported that the use of eye mask improves sleep quality, but more studies are needed to increase the quality of evidence. It is thought that transferring low-cost and easily applicable interventions that can be used to control environmental stressors such as noise and light that negatively affect sleep quality, especially in intensive care environments, into clinical practice will improve the quality of nursing care.

ELIGIBILITY:
Inclusion Criteria:

* had undergone abdominal surgery
* over 18 years of age,
* who speak Turkish,
* who have not received any diagnosis related to mental health,
* who are open to communication and co-operation
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* patients with a history of neurological or psychiatric disorders
* patients with any eye disease
* patients who are unable or unwilling to wear an eye mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Sleep status | On the 3rd postoperative day
  This form was developed by the researcher using the literature on the subject. The form was filled in based on the self-report of the patients. In order to determine the sleep status of the patients, the form included 5 statements: 'I feel tired and sleepy during the day despite sleeping for a sufficient amount of time', 'I have difficulty falling asleep 2-3 nights a week', 'I have to constantly move my legs in bed', 'I have to go to the toilet at least once during the night', 'I wake up tired and with a headache in the morning'.
Richmond Agitation Sedation Scale (RASS) Score | Postoperative 1st, 2nd and 3rd days
  It is a ten-level scale developed by Cook and Palma (1989) in which eye contact, which is not present in other scales, is evaluated following the verbal stimulus. In the scale, a score of '0' indicates the ideal level where the patient is awake and calm, while values up to '+4' reflect increasing agitation and values up to '-5' reflect increasing sedation level. As the scale score increases, it is interpreted as the agitation status of the patients worsens.
Richard-Campbell Sleep Scale (RCS) Score | Postoperative 1st, 2nd and 3rd days
  Richard-Campbell Sleep Scale (RCS): In 1987, the Turkish validity and reliability study of the scale was conducted by Richards in 2015 by Özlü and Özer. The scale consists of 6 items evaluating sleep quality, depth of sleep at night, frequency of awakening, ambient sound level, time of staying awake and time to fall asleep. Each item is evaluated on a scale ranging from 0 to 100. A score between '0-25' indicates very poor sleep and a score between '76-100' indicates very good sleep. As the scale score increases, patients' It is interpreted that sleep quality has increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Zafer Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 12 months after publication